CLINICAL TRIAL: NCT05351983
Title: Patient-derived Organoid Generation in Pancreatic Cancer: a Single Centre, Open-label, Single Arm Feasibility Study
Brief Title: Patient-derived Organoids Drug Screen in Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. med. Dres. h.c. Jan Schmidt, MME (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dres. h.c. Jan Schmidt, MME, Principal Investigator, Klinik Hirslanden, Zurich
Organization: Klinik Hirslanden, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HIRSLANDEN_PANC_001
Record Dates: First submitted 2022-04-01; First posted 2022-04-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2023-12

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm; Pancreas Adenocarcinoma; Pancreatic Cancer; Pancreatic Neoplasms; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Organoid generation (Experimental): All patients will included in a single-arm. Participants will undergo biopsy of tumor tissue for subsequent organoid generation.
  Interventions: Procedure: Surgical biopsy of tumoral tissue for organoid generation

INTERVENTIONS:
Procedure: Surgical biopsy of tumoral tissue for organoid generation — In surgically-resectable lesions, tumoral samples will be collected from the main surgical specimens, before sending it for final pathological examination. Patients with metastatic disease, will be offered to undergo port-a-cath implantation for chemotherapy delivery and concomitant laparoscopic surgical excisional biopsy of suspicious metastatic lesions. Intraoperative frozen section will confirm the presence of malignant cells in the sample. Part of the specimen will be sent for assessment of contamination by bacterial and/or fungal flora by the Microbiology Laboratory. The remaining tumour sample will be sent for patient-derived organoid (PDO) formation. Two patients' blood samples will be retrieved in ethylenediaminetetraacetic acid (EDTA) tubes and will be sent with the surgical specimen. All patients will then receive the standard of care (SOC) treatment according to the clinical judgement of the oncologist in charge, always within the framework of the international guidelines.

SUMMARY:
Few chemotherapeutic options exist for pancreatic cancer. Moreover, objective criteria are lacking for deciding which regimen is more beneficial for patient presenting with metastases at diagnosis.

This study investigates whether organoid generation from tumour samples of pancreatic cancer is a safe and feasible process for testing of multiple chemotherapy regimens in the laboratory.

By participating to this study, patients will have a part of the tumour tissue retrieved and sent to the laboratory for organoid generation and drug testing. For surgically-resectable tumors, tumoral tissue samples will be collected from the main surgical specimens, before sending it for final pathological examination. In case of suspected metastatic lesion at diagnosis, curative surgery is not indicated. Therefore, we will offer patients to undergo port-a-cath implantation for chemotherapy delivery and concomitant laparoscopic surgical excisional biopsy of suspicious metastatic (either hepatic or peritoneal) lesions.

At this stage of the study, the treatment that the patient will receive after surgery will not be affected by the results of the laboratory testing. In fact, all patients will receive the standard of care treatment based on the most recent oncologic guidelines and on the oncologist's clinical judgement. As part of the study, each patient will be followed for 30 days to assess possible surgical complications related to the surgical biopsy.

This study will help to speed up the implementation of organoid generation in the clinical routine for the choice of the best treatment of patients affected by pancreatic cancer.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent provided
* Patients older than 18 years
* Histologically- or cytologically-proven pancreatic ductal adenocarcinoma (PDAC)
* Tumour lesion amenable for laparoscopic, surgical biopsy
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0-2
* Radiologically measurable disease
* Life expectancy > 3 months
* Absolute neutrophile count >1500/microL, platelets >100'000/microL
* Serum creatinine <1.5 times of the upper limit of normal or Clearance >50ml/min (according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula)

Exclusion criteria:

* Concomitant need for full anticoagulation that cannot be interrupted or bridged prior to tissue biopsy
* ECOG PS >2
* Heart failure (NYHA class III-IV)
* Severe or uncontrolled concurrent illness
* Myocardial infarction within the previous 6 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the process | 30 days after the last patient enrollment.
  To determine the proportion of patients (specifically, the percentage with respect to the total sample enrolled in the study) for which organoids can be successfully generated and in which an effective treatment can be identified by drug screens in these patient-derived organoids. Successful generation of organoids will be defined as the presence of individual three-dimensional structures within 10 days from the begin of generation process. Effective treatment is considered a treatment decreasing of 50% (or more) the viability of patient-derived organoids.

SECONDARY OUTCOMES:
Safety of surgical biopsy and post-operative surgical complications. | 30 days post-operatively
  To evaluate safety of surgical biopsy for patient-derived organoids generation in patients with pancreatic cancer. Safety will be evaluated in terms of absolute and relative (%) number of postoperative complications. Severity will be graded according the Clavien-Dindo classification for surgical complications: complications equal to or greater than grade 3B will be considered as "severe". Management of each complication will be recorded for descriptive purposes.
Contamination rates | 30 days after the last patient enrollment.
  To assess the rate of contaminated samples by endogenous bacterial and fungal flora and to highlight possible implications in patient-derived organoid testing response.
Chemosensitivity testing | 6 days after the last organoid generation
  To assess in vitro efficacy of different chemotherapeutic regimens (and their combinations). In vitro efficacy will be evaluated based on the drug's (or drug combination's) capacity to decrease organoid viability of more than 50% after 6 days from their administration. Drugs (or their combination) tested in vitro will include Oxaliplatin, Carboplatin, Cisplatin, SN-38 (Irinotecan), Leucovorin, 5-FU, Gemcitabine, Olaparib, Nab-Paclitaxel, Nanoliposomal irinotecan (Nal-IRI), Niraparib.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Helbling, Dr. Med., Study Chair — Onkozentrum Zürich; Marianna Kruithof-De Julio, Prof. Dr. phil., Study Chair — University of Bern
Locations (1):
- Hirslanden Kliniks, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiriac H, Bucobo JC, Tzimas D, Grewel S, Lacomb JF, Rowehl LM, Nagula S, Wu M, Kim J, Sasson A, Vignesh S, Martello L, Munoz-Sagastibelza M, Somma J, Tuveson DA, Li E, Buscaglia JM. Successful creation of pancreatic cancer organoids by means of EUS-guided fine-needle biopsy sampling for personalized cancer treatment. Gastrointest Endosc. 2018 Jun;87(6):1474-1480. doi: 10.1016/j.gie.2017.12.032. Epub 2018 Jan 9. PMID 29325707
- [Background] Tiriac H, Belleau P, Engle DD, Plenker D, Deschenes A, Somerville TDD, Froeling FEM, Burkhart RA, Denroche RE, Jang GH, Miyabayashi K, Young CM, Patel H, Ma M, LaComb JF, Palmaira RLD, Javed AA, Huynh JC, Johnson M, Arora K, Robine N, Shah M, Sanghvi R, Goetz AB, Lowder CY, Martello L, Driehuis E, LeComte N, Askan G, Iacobuzio-Donahue CA, Clevers H, Wood LD, Hruban RH, Thompson E, Aguirre AJ, Wolpin BM, Sasson A, Kim J, Wu M, Bucobo JC, Allen P, Sejpal DV, Nealon W, Sullivan JD, Winter JM, Gimotty PA, Grem JL, DiMaio DJ, Buscaglia JM, Grandgenett PM, Brody JR, Hollingsworth MA, O'Kane GM, Notta F, Kim E, Crawford JM, Devoe C, Ocean A, Wolfgang CL, Yu KH, Li E, Vakoc CR, Hubert B, Fischer SE, Wilson JM, Moffitt R, Knox J, Krasnitz A, Gallinger S, Tuveson DA. Organoid Profiling Identifies Common Responders to Chemotherapy in Pancreatic Cancer. Cancer Discov. 2018 Sep;8(9):1112-1129. doi: 10.1158/2159-8290.CD-18-0349. Epub 2018 May 31. PMID 29853643
- [Background] Aung KL, Fischer SE, Denroche RE, Jang GH, Dodd A, Creighton S, Southwood B, Liang SB, Chadwick D, Zhang A, O'Kane GM, Albaba H, Moura S, Grant RC, Miller JK, Mbabaali F, Pasternack D, Lungu IM, Bartlett JMS, Ghai S, Lemire M, Holter S, Connor AA, Moffitt RA, Yeh JJ, Timms L, Krzyzanowski PM, Dhani N, Hedley D, Notta F, Wilson JM, Moore MJ, Gallinger S, Knox JJ. Genomics-Driven Precision Medicine for Advanced Pancreatic Cancer: Early Results from the COMPASS Trial. Clin Cancer Res. 2018 Mar 15;24(6):1344-1354. doi: 10.1158/1078-0432.CCR-17-2994. Epub 2017 Dec 29. PMID 29288237
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Background] Clevers H. Modeling Development and Disease with Organoids. Cell. 2016 Jun 16;165(7):1586-1597. doi: 10.1016/j.cell.2016.05.082. PMID 27315476
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Dancey JE, Dodd LE, Ford R, Kaplan R, Mooney M, Rubinstein L, Schwartz LH, Shankar L, Therasse P. Recommendations for the assessment of progression in randomised cancer treatment trials. Eur J Cancer. 2009 Jan;45(2):281-9. doi: 10.1016/j.ejca.2008.10.042. PMID 19097775
- [Background] Pazdur R. Endpoints for assessing drug activity in clinical trials. Oncologist. 2008;13 Suppl 2:19-21. doi: 10.1634/theoncologist.13-S2-19. PMID 18434634
- See also: National Comprehensive Cancer Network (NCCN) Guidelines for Pancreatic adenocarcinoma ver. 2.2021 — https://www.nccn.org/professionals/physician_gls/pdf/pancreatic.pdf